CLINICAL TRIAL: NCT01309022
Title: Immunosuppressive Medications for Previous Participants in Clinical Trial NIS01 (ITN005CT, NCT00014911)
Brief Title: Immunosuppressive Medications for Participants in ITN005CT (NCT00014911)
Status: No longer available | Type: Expanded Access
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Immune Tolerance Network (ITN) (Network)
Responsible Party: Sponsor
Other Study IDs: DAIT ITN040CT; EXIIST (Other: Immune Tolerance Network)
Record Dates: First submitted 2011-03-02; First posted 2011-03-04 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2016-02

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Diabetes Mellitus, Type 1; T1D; T1DM; Islets of Langerhans Transplantation; Pancreatic Islets Transplantation; Islet Transplant; Tacrolimus; Sirolimus; Mycophenolate mofetil; Mycophenolic acid
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Sirolimus; Tacrolimus; Mycophenolic Acid

INTERVENTIONS:
Drug: Sirolimus — Obtained by prescription and given at doses used in ClinicalTrials.gov record NCT00014911.
  Other Names: Rapamune®
Drug: Tacrolimus — Obtained by prescription and given at doses used in ClinicalTrials.gov record NCT00014911.
  Other Names: Prograf®
Drug: Mycophenolate mofetil — Obtained by prescription and given at doses used in ClinicalTrials.gov record NCT00014911.
  Other Names: MMF; CellCept
Drug: Mycophenolic acid — Obtained by prescription and given at doses used in ClinicalTrials.gov record NCT00014911.
  Other Names: Myfortic®

SUMMARY:
The purpose of this protocol is to provide continued acess to immunosuppressive medications to subjects from the completed/closed trial ITN005CT (NIS01,NCT00014911). THIS PROTOCOL DOES NOT PROVIDE MEDICINES TO DIABETES PATIENTS WHO DID NOT PARTICIPATE IN ITN005CT.

DETAILED DESCRIPTION:
Study acronym: EXIIST - Extended Immunosuppression in Islet Transplantation

Islet transplantation is an experimental therapy in people with difficult to control Type 1 diabetes (T1D). Insulin producing cells (islets) are isolated from a pancreas. After the cells are prepared, the islets are put into the subject's liver. These transplanted islets may produce insulin that the subject's islets can no longer make. In order to help keep up the function of the transplanted islets, immunosuppressive medications must be given indefinitely or for as long as the study doctor determines is necessary. The medications serve to modify the immune system that normally tries to destroy (reject) new islets.

Participants in this study have received up to three islet cell infusions as a previous participant in the ITN005CT (NIS01) protocol. They also received a maintenance immunosuppressive treatment regimen consisting of a combination of orally administered drugs (tacrolimus (Prograf®), sirolimus (Rapamune®), mycophenolate mofetil (MMF, Cellcept®), and/or mycophenolic acid (MPA, Myfortic®).) This protocol provides a way to supply these immunosuppressive medications to subjects whose islets continue to function and make C-peptide.

Routine study follow-up visits will occur on an annual and -as warranted basis.

ELIGIBILITY:
Inclusion Criteria:

* Participation in clinical trial ITN005CT (reference: ClinicalTrials.gov record NCT00014911) at Harvard University (Massachusetts General Hospital), Washington University, or University of Miami.
* Immunosuppressive regimen consisting of a single agent or some combination from among the following: tacrolimus, sirolimus, mycophenolate mofetil, and mycophenolic acid.
* Willingness of participants to use an approved method of contraception before, during, and 12 weeks after study participation.
* Peak C-peptide >0.1 pmol/mL during a mixed meal tolerance test (MMTT) within 12 months of the screening visit.

Exclusion Criteria:

* Inability to understand and sign the informed consent document for this study.
* Any medical condition which in the opinion of the investigator should preclude participation.
* Serum creatinine > 1.6 mg/dL
* Insulin requirement > 1.0 IU/kg/day
* Hemoglobin A1C (HbA1C) result > 12%
* Hypoglycemia unawareness defined as the absence of adequate autonomic symptoms at plasma glucose levels of < 54 mg/dL requiring treatment with glucagon, outside assistance, or treatment in an emergency room or hospital within a 12-month period

Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Daniel C. Brennan, MD, Study Chair — Washington University School of Medicine
Locations (3):
- United States (3):
  - University of Miami, Miami, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Washington University, St Louis, Missouri

REFERENCES:
- [Background] Shapiro AM, Ricordi C, Hering BJ, Auchincloss H, Lindblad R, Robertson RP, Secchi A, Brendel MD, Berney T, Brennan DC, Cagliero E, Alejandro R, Ryan EA, DiMercurio B, Morel P, Polonsky KS, Reems JA, Bretzel RG, Bertuzzi F, Froud T, Kandaswamy R, Sutherland DE, Eisenbarth G, Segal M, Preiksaitis J, Korbutt GS, Barton FB, Viviano L, Seyfert-Margolis V, Bluestone J, Lakey JR. International trial of the Edmonton protocol for islet transplantation. N Engl J Med. 2006 Sep 28;355(13):1318-30. doi: 10.1056/NEJMoa061267. PMID 17005949
- [Result] Brennan DC, Kopetskie HA, Sayre PH, Alejandro R, Cagliero E, Shapiro AM, Goldstein JS, DesMarais MR, Booher S, Bianchine PJ. Long-Term Follow-Up of the Edmonton Protocol of Islet Transplantation in the United States. Am J Transplant. 2016 Feb;16(2):509-17. doi: 10.1111/ajt.13458. Epub 2015 Oct 3. PMID 26433206
- See also: Immune Tolerance Network (ITN) Web Site — http://www.immunetolerance.org